CLINICAL TRIAL: NCT02114424
Title: Night Balance for Positional Obstructive Sleep Apnea Syndrome (POSAS) A Prospective, Randomized, Controlled Open Trial in Daily Clinical Practice
Brief Title: Night Balance for Positional Obstructive Sleep Apnea Syndrome (POSAS)
Acronym: POSAS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Philip Tønnesen, M.D., Senior consultant, Dept. of Sleep, Dept. of Clin. neurophysiology, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-3-2014-039
Record Dates: First submitted 2014-04-10; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Obstructive Sleep Apnea (OSAS)
Keywords: Positional Obstructive sleep apnea syndrome (POSAS); Obstructive sleep apnea syndrome (OSAS); Apnea-Hypnea Index (AHI); Sleep questionnaire; Positional sleep apnea belt; Adverse events; Compliance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positional vibrator belt (Active Comparator): Positional belt to avoid supine sleep.
  Interventions: Device: Positional vibrator belt
- No Night balance (No Intervention): the first 2 months without Night Balance

INTERVENTIONS:
Device: Positional vibrator belt — Belt with vibarator to avoid sleep supine
  Other Names: Night Balance, B.V,, 2629 JD Delft, The Netherlands
  Arms: Positional vibrator belt

SUMMARY:
POSAS can be treated with CPAP however there is now evidence from a few studies that Night Balance is effective in POSAS. Night Balance seems to be better accepted than CPAP so we would like to examine if we could find similar results in routine clinical work and especially we would like to confirm the subjective effects with objective measures i.e. a reduction in AHI in the supine position during sleep.

DETAILED DESCRIPTION:
Primary aim: Efficacy and adherence of Night Balance in POSAS versus no therapy after 2 months (Sleep supine).

Secondary aim: Efficacy and adherence of Night Balance in POSAS after a 6 months period (Sleep supine and compliance and AHI).

Nigh Balance is a vibrator and a belt that vibrate when laying supine so that after a few days you will not sleep supine.

ELIGIBILITY:
Inclusion Criteria:

* AHI supine ≥ AHI non-supine x 2,
* AHI supine ≥ 10
* AHI non-supine <10
* 10 -90 % sleep time in supine position
* Daytime tiredness and/or disturbed sleep and/or snoring

Exclusion Criteria:

* Not able or willing to cooperate
* Age <18 years
* Central Sleep Apnea
* Night or shifting work
* Severe chronic heart failure or severe COPD
* A medical history of known causes of tiredness by day or severe sleep disruption (insomnia, PLMS, Narcolepsy)
* Seizure disorder
* A known medical history of mental retardation, memory disorders or psychiatric disorders
* The inability to provide informed consent
* Pacemaker
* Pain in joints or shoulder
* Other reasons unable to sleep in lateral positions.
* Pregnant females or females that plan pregnancy in study period (problems sleeping supine)
* Breastfeeding females in study period (other reasons for disturbed sleep)
* Plan weight reduction in study period
* Plan to quit smoking in study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-06 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy and adherence of Night Balance in POSAS versus no therapy after 2 months (Sleep supine and AHI). | After 2 months
  AFter 2 months assessment will be done by sleep questionnaires and CRM

SECONDARY OUTCOMES:
Efficacy and adherence of Night Balance in POSAS versus no therapy after 2 months (Sleep supine). | 6 months after entry
  ALl wil ahve a new CRM after 6 months with Night Balance and sleep questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Philip Toennesen, M.D., Ph.D., Principal Investigator — GlsotrupUH
Locations (1):
- Glostrup University Hospital, Glostrup Municipality, Denmark

REFERENCES:
- [Background] 23. van der Star A, Mekking S, van Riet M. The technical validation of the Sleep Position Trainer. Nightbalance Research and Development [Internet]. 2012 Oct [cited 2013 Dec 6]:1-12. Available from http://www.nightbalance.com/research.